CLINICAL TRIAL: NCT02181790
Title: Addition of 308-nm Excimer Laser to Acitretin Therapy in the Management of Palmoplantar Psoriasis
Brief Title: Addition of Excimer Laser to Treatment With Acitretin Tablets for Psoriasis of the Palms and Soles
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of subjects
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mark Lebwohl, Professor & Chair Dermatology, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-0580; PD14-01323 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis, Skin or Nails
Keywords: psoriasis; palmoplantar; acitretin; retinoids; laser treatment
MeSH Terms: conditions — Psoriasis | interventions — Lasers, Excimer; Laser Therapy; Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Group (Experimental): excimer laser treatment to one palm and/or one sole
  Interventions: Device: Excimer laser; Drug: Acitretin
- Second Group (Experimental): excimer laser treatment to both palms and/or soles
  Interventions: Device: Excimer laser; Drug: Acitretin

INTERVENTIONS:
Device: Excimer laser — twice weekly treatments with the excimer laser for a total of 8 weeks.
  Other Names: laser treatment
Drug: Acitretin — 17.5mg/d
  Other Names: Soriatane

SUMMARY:
Psoriasis is a common skin disease that can affect 1-3% of the population. For more severe psoriasis, oral medication such as acitretin is sometimes given. While acitretin may be sufficient for treatment of some patients, psoriasis of the palms and soles is particularly challenging to treat, and may not respond to acitretin alone.

In this study, the focus is on patients who have psoriasis of the palms and soles, and are currently taking acitretin. The aim is to initially recruit 10 patients and offer them treatment with a laser, the excimer laser, to one palm and one sole. Patients will receive laser treatment twice weekly for a total of 8 weeks, while also taking their acitretin tablet. If the side treated with the excimer laser shows greater improvement compared to the other side, the second part of the study will be conducted.

In this second part, another 15 patients will be included. These patients will receive twice weekly treatments with the excimer laser to one both palms and/or soles, for a total of 8 weeks. The aim is to prove that the addition of excimer laser to treatment with acitretin will lead to greater improvement of psoriasis on palms and soles.

DETAILED DESCRIPTION:
This open label study evaluated whether a reduction in acitretin dose from 25 mg/day to 17.5 mg/day in patients with severe plaque-type psoriasis undergoing phototherapy treatment improved tolerability while maintaining comparable efficacy.

At baseline, subjects were switched from 25 to 17.5 mg acitretin daily and followed for 12 weeks.

Efficacy evaluations were performed through week 12. The psoriasis area-and severity index (termed PASI) combines assessments of the extent of body-surface involvement in four anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration (thickness) in each region, yielding an overall score of 0 (no psoriasis) to 72 (severe disease). The physician's global assessment rates the patient's psoriasis overall relative to baseline as 1 (clear), 2 (excellent), 3 (good), 4 (fair), 5 (poor), or 6 (worse) and considers involvement of body surface area (BSA), induration, scaling, and erythema. The 10-item Dermatology Life Quality Index questionnaire, completed by the subject, measures whether psoriasis has an effect on the subject's quality of life, with scores ranging from 0 ("no effect") to 30 ("extremely large effect"). The 15-item Psoriasis Disability Index (PDI), completed by the subject, measures the level of impairment psoriasis has on quality of life, with scores ranging from 0 ("no effect") to 45 ("extremely impaired"). Subjects also completed a subjective assessment of efficacy of the reduced dose of acitretin at week 12 of the study by answering the question "How was your psoriasis over the last 3 months?", with answers ranging from better than before, the same as before, or worse than before.

The safety and tolerability was assessed for the reduced acitretin dose by monitoring adverse events and routine laboratory values through week 12. Serum samples collected at baseline and week 12 were tested for LFTs, lipids, CBC, and chemistry panel. Subjects also completed a subjective assessment of tolerability of the lower dose at week 12 of the study by answering the question, "Did your symptoms from the medicine you noted above improve over the last 3 months?", with answers ranging from better than before, the same as before, or worse than before.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age
* Diagnosis of psoriasis, with palmoplantar involvement
* Initiated on oral acitretin for treatment of their psoriasis by their physician

Exclusion Criteria:

* Subjects less than 18 years old
* Subjects with any skin disease, disease state, or physical condition that would impair evaluation of the skin
* Additional systemic therapy for psoriasis in last 4 weeks
* Additional topical or photo-therapy in last 2 weeks
* Usage of any additional therapy except for emollients and keratolytic agents (5% salicylic acid ointment or 30% urea cream)
* Pre-existent or current cutaneous malignancy affecting the palms and/or soles
* History of photosensitive disorders
* Ingestion of drugs reported to cause photosensitivity reactions
* Presence of erythroderma or generalized pustular psoriasis
* Concomitant use of sunlamps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Excimer Laser (One Palm/Sole): excimer laser treatment to one palm and/or one sole
  Excimer laser: twice weekly treatments with the excimer laser for a total of 8 weeks.
- Excimer Laser (Both Palms/Soles): excimer laser treatment to both palms and/or soles
  Excimer laser: twice weekly treatments with the excimer laser for a total of 8 weeks.
Period: Overall Study
Arm/Group | Excimer Laser (One Palm/Sole) | Excimer Laser (Both Palms/Soles)
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — study terminated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Group | Second Group | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI)
Description: The percentage of patients achieving a 75% reduction in the Psoriasis Area and Severity Index (PASI) from baseline after 16 treatments with the excimer laser in the first phase of the study.
Time Frame: baseline and week 12
Population: study terminated before study completion, no data collected
Arm/Group | First Group | Second Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Dermatology Life Quality Index (DLQI) at Week 8 From Baseline
Description: reduction in DLQI from baseline after 16 treatments with the excimer laser in the first phase of the study
Time Frame: baseline and week 8
Population: study terminated before study completion, no data collected
Arm/Group | Excimer Laser (One Palm/Sole) | Excimer Laser (Both Palms/Soles)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | First Group | Second Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No